CLINICAL TRIAL: NCT02096211
Title: 36mm CERAMAX® Ceramic Hip System PMA PAS STUDY: Short to Mid-Term Follow-up , New Study Subjects (Ceramic Hip System, Subjects Receive CERAMAX 36mm Ceramic Acetabular Bearing Insert That Articulates With a Ceramic Femoral Head for THA)
Brief Title: Ceramic-on-Ceramic (COC) 36mm Acetabular Bearing Insert Post Approval Study-New Subjects (COC36mmPAS)
Acronym: COC36mmPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12017
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Results first posted 2025-05-06 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Non-inflammatory Degenerative Joint Disease; Osteoarthritis; Avascular Necrosis; Post-Traumatic Osteoarthritis of Hip
Keywords: Total hip replacement; Total hip arthroplasty; Hip joint replacement; Hip prosthesis replacement
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CERAMAX COC 36mm Acetabular Cup (Other): The CERAMAX 36mm ceramic acetabular bearing insert component is manufactured from high purity, dense alumina matrix composite ceramic.The insert is available in several inner diameter sizes, including 36mm; only 36mm inserts will be utilized in this PAS. The inserts secure to DePuy's Pinnacle acetabular shells by means of an interlocking mechanical taper.
  Interventions: Device: COC 36mm

INTERVENTIONS:
Device: COC 36mm — Total Hip Replacement with COC 36mm Acetabular Cup System
  Other Names: CERAMAX; CERAMAX 36mm; CERAMAX Acetabular System; 36mm CERAMAX Acetabular System

SUMMARY:
This study is intended to gather short (Pre-operative to 4-years) and mid-term (5-years) information regarding the performance and safety of the commercially available 36mm CERAMAX® Ceramic on Ceramic Total Hip System from a cohort of new study subjects that were not previously involved in the IDE study for this device.

DETAILED DESCRIPTION:
Up to 10 (up to 5 original IDE + 5 new sites)

A prospective, non-controlled, non-randomized, multicenter study. Subjects will be seen for a clinic visit pre-operatively at the time of consent, (-90 days to surgery) and then at post-operatively at 6 weeks (1-92 days), 1 year (275-455 days), 2 years (640-820 days) and 3 years (1005-1185days), 4 years (1370-1550 days), and a minimum of 5 years (1825- 2555 days).

Data collected will include: Pre-operatively subject history and demographics; Operative and device details; and Post-operatively Harris HIp scores, Subject Hip Outcomes, and Adverse Events.

In order to optimize mid-term follow-up compliance, site personnel are permitted to contact the study subject in the 3 and 4 year intervals by phone (in place of a clinic visit) to assess the current status of the hip.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 21 - 75 at the time of surgery.
* Individuals, who in the opinion of the investigator, are suitable candidates for primary total hip replacement using the devices specified in this protocol.
* Individuals with non-inflammatory degenerative joint disease (NIDJD) or any of its composite diagnoses of osteoarthritis, avascular necrosis, and posttraumatic arthritis.
* Individuals who are willing and able to provide informed patient consent for participation in the study;
* Individuals who are willing and able to return for follow-up as specified by the study protocol; and
* Individuals who are willing and able to complete the Subject Hip Outcomes questionnaire as specified by the study protocol.

Exclusion Criteria:

* Skeletally immature patients (tibial and femoral epiphyses not closed)
* Evidence of active infections that may spread to other areas of the body (e.g.,osteomyelitis, pyogenic infection of the hip joint, overt infection, urinary tract infection, etc.)
* The presence of any known neoplastic (tumor-causing) or metastatic (spread of cancerous cells) disease
* Significant neurologic or musculoskeletal disorders or diseases that may adversely affect gait, weight bearing or postoperative recovery (e.g., muscular dystrophy, multiple sclerosis)
* Presence of highly communicable disease(s) that may limit follow-up (e.g., immuno-compromised conditions, hepatitis, active tuberculosis, etc.)
* Any condition that may interfere with postoperative recovery (e.g., Paget's disease, Charcot's disease)
* Inadequate bone stock to support the device (e.g., severe osteopenia orosteoporosis)
* Poor skin coverage around the hip joint
* Use in patients with known allergies to the implant materials
* Marked atrophy (muscle and/or tissue loss) or deformity in the upper femur such as a birth defect affecting the leg bones.
* Inflammatory degenerative joint disease (like rheumatoid arthritis)
* Subject has participated in an IDE/IND clinical investigation, other than the COC28/COC36 IDE or PAS for their contralateral hip, with an investigational product in the last three months.
* Subject is currently involved in a personal injury litigation, medical-legal or worker's compensation claims.
* Subject is a known drug or alcohol abuser or has a psychological disorder that could affect their ability to comply with protocol procedures and/or subject-completed questionnaires.
* The Subject is a woman who is pregnant or lactating.
* The Subject has a medical condition with less than 2 years of life expectancy.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terrence D Whalen, BS, DC, Study Director — DePuy Orthopaedics
Locations (13):
- United States (9):
  - Joint Surgeons of Sacremento, Sacramento, California
  - Colorado Joint Replacement, Denver, Colorado
  - Florida Orthopaedic Institute, Tampa, Florida
  - Arthroplasty Foundation, Louisville, Kentucky
  - TUFTS - New England Medical Center, Boston, Massachusetts
  - New England Baptist Hospital, Boston, Massachusetts
  - Samuel Wellman, MD / Duke University Medical Center, Durham, North Carolina
  - Orthopedic One, Columbus, Ohio
  - UPenn, Philadelphia, Pennsylvania
- Canada (4):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Queens University - Kingston General Hospital, Kingston, Quebec
  - McGill University - Jewish General Hospital, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All eligible patients were asked if they were interested in study participation
Units Other Than Participants: Implants
Period: Overall Study
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Started | 170; 172 Implants
Completed | 110; 110 Implants
Not Completed | 60; 62 Implants
Not completed — Death | 2
Not completed — Withdrawal by Subject | 8
Not completed — Revision of implant | 7
Not completed — Lost to Follow-up | 43

BASELINE CHARACTERISTICS:
Population: All study Participants (n=170)
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 170
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in years of study participants (n=170) Population: All study participants (n=170)
  Years
    Participant Age | 53.6 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants] — Participant gender (n=170) Population: Study Participant Gender
  Participants
    Female | 70
    Male | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Study Participant Ethnicity Population: Study Participants
  Participants
    Study Participant Ethnicity: Hispanic or Latino | 2
    Study Participant Ethnicity: Not Hispanic or Latino | 168
    Study Participant Ethnicity: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Study Participant Race Population: Study Participants
  Participants
    Study Participant Race: American Indian or Alaska Native | 1
    Study Participant Race: Asian | 0
    Study Participant Race: Native Hawaiian or Other Pacific Islander | 0
    Study Participant Race: Black or African American | 26
    Study Participant Race: White | 143
    Study Participant Race: More than one race | 0
    Study Participant Race: Unknown or Not Reported | 0
Study Participant Primary Diagnosis [Count of Participants; unit: Participants] — Study Participant Primary Diagnosis Population: Study Participants
  Participants
    Osteoarthritis | 144
    Avascular Necrosis | 22
    Post Traumatic Arthritis | 4

OUTCOME MEASURES:

1. Primary Outcome: Post-Operative 5-Year Device Survivorship
Description: Device survivorship at 5 years post-operatively was the primary endpoint in this study. A revision is defined as the removal of any Total Hip Arthroplasty (THA) component(s), and device survival is defined as the lack of revision. A 5-year Kaplan-Meier survivorship estimate of COC 36 mm implanted hips is provided.
Time Frame: 5 years
Population: All Study Participants
Measure: Number (95% Confidence Interval); unit: Percentage of implants
Units Other Than Participants: Implants
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 170
Number analyzed (Implants) | 172
Percentage of implants | 95.3 [90.8 to 97.6]

2. Secondary Outcome: Kaplan Meier Device Survivorship at Years 1 Through 6
Description: Device survivorship at each year post-operative was a secondary endpoint in this study. A revision is defined as the removal of any Total Hip Arthroplasty (THA) component(s), and device survival is defined as the lack of revision. A Kaplan-Meier survivorship estimate of COC 36 mm implanted hips is provided for each post-operative year.
Time Frame: Years 1 through 6 post-operatively
Population: All study participants
Measure: Number (95% Confidence Interval); unit: Percentage of implants
Units Other Than Participants: Implants
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 170
Number analyzed (Implants) | 172
Percentage of implants
  Kaplan Meier device survivorship at 1 year with 164 hips remaining: number analyzed (Participants) | 164
  Kaplan Meier device survivorship at 1 year with 164 hips remaining: number analyzed (Implants) | 164
  Kaplan Meier device survivorship at 1 year with 164 hips remaining | 97.7 [93.9 to 99.1]
  Kaplan Meier device survivorship at 2 years with 161 hips remaining: number analyzed (Participants) | 161
  Kaplan Meier device survivorship at 2 years with 161 hips remaining: number analyzed (Implants) | 161
  Kaplan Meier device survivorship at 2 years with 161 hips remaining | 96.5 [92.3 to 98.4]
  Kaplan Meier device survivorship at 3 years with 158 hips remaining: number analyzed (Participants) | 158
  Kaplan Meier device survivorship at 3 years with 158 hips remaining: number analyzed (Implants) | 158
  Kaplan Meier device survivorship at 3 years with 158 hips remaining | 95.9 [91.6 to 98.0]
  Kaplan Meier device survivorship at 4 years with 154 hips remaining: number analyzed (Participants) | 154
  Kaplan Meier device survivorship at 4 years with 154 hips remaining: number analyzed (Implants) | 154
  Kaplan Meier device survivorship at 4 years with 154 hips remaining | 95.3 [90.8 to 97.6]
  Kaplan Meier device survivorship at 5 years with 150 hips remaining: number analyzed (Participants) | 150
  Kaplan Meier device survivorship at 5 years with 150 hips remaining: number analyzed (Implants) | 150
  Kaplan Meier device survivorship at 5 years with 150 hips remaining | 95.3 [90.8 to 97.6]
  Kaplan Meier device survivorship at 6 years with 58 hips remaining: number analyzed (Participants) | 58
  Kaplan Meier device survivorship at 6 years with 58 hips remaining: number analyzed (Implants) | 58
  Kaplan Meier device survivorship at 6 years with 58 hips remaining | 95.3 [90.8 to 97.6]

3. Secondary Outcome: Annual Total Harris Hip Score
Description: The Harris Hip Score (HHS) is a standardized tool used to evaluate hip pain, function, and mobility. The HHS is score from 0 to 100, with higher scores indicating better outcomes. A score of less than 70 is considered poor, 70-80 is fair, 80-90 is good, 90-100 is excellent
Time Frame: Annually through 5 years
Population: All study participants who attended their annual clinical evaluation
Measure: Count of Units; unit: Participant hips
Units Other Than Participants: Participant hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 128
Number analyzed (Participant hips) | 128
Participant hips
  Harris Hip score at 1 year Number of participants with Excellent Scores (90-100) | 98 [lower limit 12.18]
  Harris Hip score at 1 year Number of participants with Good Scores (80-89) | 18
  Harris Hip score at 1 year Number of participants with Fair Scores (70-79) | 4
  Harris Hip score at 1 year Number of participants with Poor Scores (Less than 70) | 8
  Harris Hip score at 2 years. Number of participants with Excellent Scores (90-100): number analyzed (Participants) | 123
  Harris Hip score at 2 years. Number of participants with Excellent Scores (90-100): number analyzed (Participant hips) | 123
  Harris Hip score at 2 years. Number of participants with Excellent Scores (90-100) | 90
  Harris Hip score at 2 years. Number of participants with Good Scores (80-89): number analyzed (Participants) | 123
  Harris Hip score at 2 years. Number of participants with Good Scores (80-89): number analyzed (Participant hips) | 123
  Harris Hip score at 2 years. Number of participants with Good Scores (80-89) | 20
  Harris Hip score at 2 years. Number of participants with Fair Scores (70-79): number analyzed (Participants) | 123
  Harris Hip score at 2 years. Number of participants with Fair Scores (70-79): number analyzed (Participant hips) | 123
  Harris Hip score at 2 years. Number of participants with Fair Scores (70-79) | 6
  Harris Hip score at 2 years. Number of participants with Poor Scores (Less than 70): number analyzed (Participants) | 123
  Harris Hip score at 2 years. Number of participants with Poor Scores (Less than 70): number analyzed (Participant hips) | 123
  Harris Hip score at 2 years. Number of participants with Poor Scores (Less than 70) | 7
  Harris Hip score at 3 years. Number of participants with Excellent Scores (90-100): number analyzed (Participants) | 63
  Harris Hip score at 3 years. Number of participants with Excellent Scores (90-100): number analyzed (Participant hips) | 63
  Harris Hip score at 3 years. Number of participants with Excellent Scores (90-100) | 50
  Harris Hip score at 3 years. Number of participants with Good Scores (80-89): number analyzed (Participants) | 63
  Harris Hip score at 3 years. Number of participants with Good Scores (80-89): number analyzed (Participant hips) | 63
  Harris Hip score at 3 years. Number of participants with Good Scores (80-89) | 5
  Harris Hip score at 3 years. Number of participants with Fair Scores (70-79): number analyzed (Participants) | 63
  Harris Hip score at 3 years. Number of participants with Fair Scores (70-79): number analyzed (Participant hips) | 63
  Harris Hip score at 3 years. Number of participants with Fair Scores (70-79) | 2
  Harris Hip score at 3 years. Number of participants with Poor Scores (Less than 70): number analyzed (Participants) | 63
  Harris Hip score at 3 years. Number of participants with Poor Scores (Less than 70): number analyzed (Participant hips) | 63
  Harris Hip score at 3 years. Number of participants with Poor Scores (Less than 70) | 6
  Harris Hip score at 4 years. Number of participants with Excellent Scores (90-100): number analyzed (Participants) | 31
  Harris Hip score at 4 years. Number of participants with Excellent Scores (90-100): number analyzed (Participant hips) | 31
  Harris Hip score at 4 years. Number of participants with Excellent Scores (90-100) | 20
  Harris Hip score at 4 years. Number of participants with Good Scores (80-89): number analyzed (Participants) | 31
  Harris Hip score at 4 years. Number of participants with Good Scores (80-89): number analyzed (Participant hips) | 31
  Harris Hip score at 4 years. Number of participants with Good Scores (80-89) | 7
  Harris Hip score at 4 years. Number of participants with Fair Scores (70-79): number analyzed (Participants) | 31
  Harris Hip score at 4 years. Number of participants with Fair Scores (70-79): number analyzed (Participant hips) | 31
  Harris Hip score at 4 years. Number of participants with Fair Scores (70-79) | 1
  Harris Hip score at 4 years. Number of participants with Poor Scores (Less than 70): number analyzed (Participants) | 31
  Harris Hip score at 4 years. Number of participants with Poor Scores (Less than 70): number analyzed (Participant hips) | 31
  Harris Hip score at 4 years. Number of participants with Poor Scores (Less than 70) | 3
  Harris Hip score at 5 years. Number of participants with Excellent Scores (90-100): number analyzed (Participants) | 109
  Harris Hip score at 5 years. Number of participants with Excellent Scores (90-100): number analyzed (Participant hips) | 109
  Harris Hip score at 5 years. Number of participants with Excellent Scores (90-100) | 85
  Harris Hip score at 5 years. Number of participants with Good Scores (80-89): number analyzed (Participants) | 109
  Harris Hip score at 5 years. Number of participants with Good Scores (80-89): number analyzed (Participant hips) | 109
  Harris Hip score at 5 years. Number of participants with Good Scores (80-89) | 11
  Harris Hip score at 5 years. Number of participants with Fair Scores (70-79): number analyzed (Participants) | 109
  Harris Hip score at 5 years. Number of participants with Fair Scores (70-79): number analyzed (Participant hips) | 109
  Harris Hip score at 5 years. Number of participants with Fair Scores (70-79) | 8
  Harris Hip score at 5 years. Number of participants with Poor Scores (Less than 70): number analyzed (Participants) | 109
  Harris Hip score at 5 years. Number of participants with Poor Scores (Less than 70): number analyzed (Participant hips) | 109
  Harris Hip score at 5 years. Number of participants with Poor Scores (Less than 70) | 5

4. Secondary Outcome: Annual Harris Hip Pain Sub Score
Description: The Harris Hip Score (HHS) is a standardized tool used to evaluate hip pain, function, and mobility. The HHS is score from 0 to 100, with higher scores indicating better outcomes. A score of less than 70 is considered poor, 70-80 is fair, 80-90 is good, 90-100 is excellent
  This Secondary Outcome reports on the Pain Sub Score which has categories of None (44 points), Slight (40), Mild (30), Moderate (20), Marked (10), and Totally Disabled (0)
Time Frame: Annually through 5 years
Population: All study participants who attended their annual clinical evaluation
Measure: Count of Units; unit: Participant hips
Units Other Than Participants: Participant hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 128
Number analyzed (Participant hips) | 128
Participant hips
  Harris Hip Pain Sub Score at 1 year Participants with a "None" Score (44) | 84
  Harris Hip Pain Sub Score at 1 year Participants with a "Slight" Score (40) | 28
  Harris Hip Pain Sub Score at 1 year Participants with a "Mild" Score (30) | 7
  Harris Hip Pain Sub Score at 1 year Participants with a "Moderate" Score (20) | 6
  Harris Hip Pain Sub Score at 1 year Participants with a "Marked" Score (10) | 2
  Harris Hip Pain Sub Score at 1 year Participants with a "Totally Disabled" Score (0) | 1
  Harris Hip Pain Sub Score at 2 years Participants with a "None" Score (44): number analyzed (Participants) | 123
  Harris Hip Pain Sub Score at 2 years Participants with a "None" Score (44): number analyzed (Participant hips) | 123
  Harris Hip Pain Sub Score at 2 years Participants with a "None" Score (44) | 87
  Harris Hip Pain Sub Score at 2 years Participants with a "Slight" Score (40): number analyzed (Participants) | 123
  Harris Hip Pain Sub Score at 2 years Participants with a "Slight" Score (40): number analyzed (Participant hips) | 123
  Harris Hip Pain Sub Score at 2 years Participants with a "Slight" Score (40) | 18
  Harris Hip Pain Sub Score at 2 years Participants with a "Mild" Score (30): number analyzed (Participants) | 123
  Harris Hip Pain Sub Score at 2 years Participants with a "Mild" Score (30): number analyzed (Participant hips) | 123
  Harris Hip Pain Sub Score at 2 years Participants with a "Mild" Score (30) | 11
  Harris Hip Pain Sub Score at 2 years Participants with a "Moderate" Score (20): number analyzed (Participants) | 123
  Harris Hip Pain Sub Score at 2 years Participants with a "Moderate" Score (20): number analyzed (Participant hips) | 123
  Harris Hip Pain Sub Score at 2 years Participants with a "Moderate" Score (20) | 5
  Harris Hip Pain Sub Score at 2 years Participants with a "Marked" Score (10): number analyzed (Participants) | 123
  Harris Hip Pain Sub Score at 2 years Participants with a "Marked" Score (10): number analyzed (Participant hips) | 123
  Harris Hip Pain Sub Score at 2 years Participants with a "Marked" Score (10) | 1
  Harris Hip Pain Sub Score at 2 years Participants with a "Totally Disabled" Score (0): number analyzed (Participants) | 123
  Harris Hip Pain Sub Score at 2 years Participants with a "Totally Disabled" Score (0): number analyzed (Participant hips) | 123
  Harris Hip Pain Sub Score at 2 years Participants with a "Totally Disabled" Score (0) | 1
  Harris Hip Pain Sub Score at 3 years Participants with a "None" Score (44): number analyzed (Participants) | 67
  Harris Hip Pain Sub Score at 3 years Participants with a "None" Score (44): number analyzed (Participant hips) | 67
  Harris Hip Pain Sub Score at 3 years Participants with a "None" Score (44) | 51
  Harris Hip Pain Sub Score at 3 years Participants with a "Slight" Score (40): number analyzed (Participants) | 67
  Harris Hip Pain Sub Score at 3 years Participants with a "Slight" Score (40): number analyzed (Participant hips) | 67
  Harris Hip Pain Sub Score at 3 years Participants with a "Slight" Score (40) | 8
  Harris Hip Pain Sub Score at 3 years Participants with a "Mild" Score (30): number analyzed (Participants) | 67
  Harris Hip Pain Sub Score at 3 years Participants with a "Mild" Score (30): number analyzed (Participant hips) | 67
  Harris Hip Pain Sub Score at 3 years Participants with a "Mild" Score (30) | 2
  Harris Hip Pain Sub Score at 3 years Participants with a "Moderate" Score (20): number analyzed (Participants) | 67
  Harris Hip Pain Sub Score at 3 years Participants with a "Moderate" Score (20): number analyzed (Participant hips) | 67
  Harris Hip Pain Sub Score at 3 years Participants with a "Moderate" Score (20) | 2
  Harris Hip Pain Sub Score at 3 years Participants with a "Marked" Score (10): number analyzed (Participants) | 67
  Harris Hip Pain Sub Score at 3 years Participants with a "Marked" Score (10): number analyzed (Participant hips) | 67
  Harris Hip Pain Sub Score at 3 years Participants with a "Marked" Score (10) | 1
  Harris Hip Pain Sub Score at 3 years Participants with a "Totally Disabled" Score (0): number analyzed (Participants) | 67
  Harris Hip Pain Sub Score at 3 years Participants with a "Totally Disabled" Score (0): number analyzed (Participant hips) | 67
  Harris Hip Pain Sub Score at 3 years Participants with a "Totally Disabled" Score (0) | 0
  Harris Hip Pain Sub Score at 4 years Participants with a "None" Score (44): number analyzed (Participants) | 35
  Harris Hip Pain Sub Score at 4 years Participants with a "None" Score (44): number analyzed (Participant hips) | 35
  Harris Hip Pain Sub Score at 4 years Participants with a "None" Score (44) | 23
  Harris Hip Pain Sub Score at 4 years Participants with a "Slight" Score (40): number analyzed (Participants) | 35
  Harris Hip Pain Sub Score at 4 years Participants with a "Slight" Score (40): number analyzed (Participant hips) | 35
  Harris Hip Pain Sub Score at 4 years Participants with a "Slight" Score (40) | 6
  Harris Hip Pain Sub Score at 4 years Participants with a "Mild" Score (30): number analyzed (Participants) | 35
  Harris Hip Pain Sub Score at 4 years Participants with a "Mild" Score (30): number analyzed (Participant hips) | 35
  Harris Hip Pain Sub Score at 4 years Participants with a "Mild" Score (30) | 2
  Harris Hip Pain Sub Score at 4 years Participants with a "Moderate" Score (20): number analyzed (Participants) | 35
  Harris Hip Pain Sub Score at 4 years Participants with a "Moderate" Score (20): number analyzed (Participant hips) | 35
  Harris Hip Pain Sub Score at 4 years Participants with a "Moderate" Score (20) | 2
  Harris Hip Pain Sub Score at 4 years Participants with a "Marked" Score (10): number analyzed (Participants) | 35
  Harris Hip Pain Sub Score at 4 years Participants with a "Marked" Score (10): number analyzed (Participant hips) | 35
  Harris Hip Pain Sub Score at 4 years Participants with a "Marked" Score (10) | 2
  Harris Hip Pain Sub Score at 4 years Participants with a "Totally Disabled" Score (0): number analyzed (Participants) | 35
  Harris Hip Pain Sub Score at 4 years Participants with a "Totally Disabled" Score (0): number analyzed (Participant hips) | 35
  Harris Hip Pain Sub Score at 4 years Participants with a "Totally Disabled" Score (0) | 0
  Harris Hip Pain Sub Score at 5 years Participants with a "None" Score (44): number analyzed (Participants) | 110
  Harris Hip Pain Sub Score at 5 years Participants with a "None" Score (44): number analyzed (Participant hips) | 110
  Harris Hip Pain Sub Score at 5 years Participants with a "None" Score (44) | 81
  Harris Hip Pain Sub Score at 5 years Participants with a "Slight" Score (40): number analyzed (Participants) | 110
  Harris Hip Pain Sub Score at 5 years Participants with a "Slight" Score (40): number analyzed (Participant hips) | 110
  Harris Hip Pain Sub Score at 5 years Participants with a "Slight" Score (40) | 15
  Harris Hip Pain Sub Score at 5 years Participants with a "Mild" Score (30): number analyzed (Participants) | 110
  Harris Hip Pain Sub Score at 5 years Participants with a "Mild" Score (30): number analyzed (Participant hips) | 110
  Harris Hip Pain Sub Score at 5 years Participants with a "Mild" Score (30) | 7
  Harris Hip Pain Sub Score at 5 years Participants with a "Moderate" Score (20): number analyzed (Participants) | 110
  Harris Hip Pain Sub Score at 5 years Participants with a "Moderate" Score (20): number analyzed (Participant hips) | 110
  Harris Hip Pain Sub Score at 5 years Participants with a "Moderate" Score (20) | 7
  Harris Hip Pain Sub Score at 5 years Participants with a "Marked" Score (10): number analyzed (Participants) | 110
  Harris Hip Pain Sub Score at 5 years Participants with a "Marked" Score (10): number analyzed (Participant hips) | 110
  Harris Hip Pain Sub Score at 5 years Participants with a "Marked" Score (10) | 0
  Harris Hip Pain Sub Score at 5 years Participants with a "Totally Disabled" Score (0): number analyzed (Participants) | 110
  Harris Hip Pain Sub Score at 5 years Participants with a "Totally Disabled" Score (0): number analyzed (Participant hips) | 110
  Harris Hip Pain Sub Score at 5 years Participants with a "Totally Disabled" Score (0) | 0

5. Secondary Outcome: Annual Harris Hip Function and Activity Score
Description: The Harris Hip Score (HHS) is a standardized tool used to evaluate hip pain, function, and mobility. The HHS is score from 0 to 100, with higher scores indicating better outcomes. A score of less than 70 is considered poor, 70-80 is fair, 80-90 is good, 90-100 is excellent
  This Secondary Outcome reports on the Function and Activity Sub Score which has categories of Normal (40-47 points), Mild Dysfunction (30-39), Moderate Dysfunction (20-29), Severe Dysfunction (10-19), and Disabled (0 - 9)
Time Frame: Annually through 5 years
Population: All Study Participants who attended their annual clinical evaluation
Measure: Count of Units; unit: Participant Hips
Units Other Than Participants: Participant Hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 128
Number analyzed (Participant Hips) | 128
Participant Hips
  Harris Hip Function and Activity Score at 1 Year Subjects with a "Normal" Score (40-47) | 96
  Harris Hip Function and Activity Score at 1 Year Subjects with a "Mild Dysfunction" Score (30-39) | 28
  Harris Hip Function and Activity Score at 1 Yr Subjects with a "Moderate Dysfunction" Score (20-29) | 3
  Harris Hip Function and Activity Score at 1 Year Subjects with a "Severe Dysfunction" Score (10-19) | 1
  Harris Hip Function and Activity Score at 1 Year Subjects with a "Disabled" Score (0-9) | 0
  Harris Hip Function and Activity Score at 2 Years Subjects with a "Normal" Score (40-47): number analyzed (Participants) | 123
  Harris Hip Function and Activity Score at 2 Years Subjects with a "Normal" Score (40-47): number analyzed (Participant Hips) | 123
  Harris Hip Function and Activity Score at 2 Years Subjects with a "Normal" Score (40-47) | 99
  Harris Hip Function and Activity Score at 2 Years Subjects with a "Mild Dysfunction" Score (30-39): number analyzed (Participants) | 123
  Harris Hip Function and Activity Score at 2 Years Subjects with a "Mild Dysfunction" Score (30-39): number analyzed (Participant Hips) | 123
  Harris Hip Function and Activity Score at 2 Years Subjects with a "Mild Dysfunction" Score (30-39) | 16
  Harris Hip Function and Activity Score at 2 Yrs Subjects with a "Moderate Dysfunction" Score (20-29): number analyzed (Participants) | 123
  Harris Hip Function and Activity Score at 2 Yrs Subjects with a "Moderate Dysfunction" Score (20-29): number analyzed (Participant Hips) | 123
  Harris Hip Function and Activity Score at 2 Yrs Subjects with a "Moderate Dysfunction" Score (20-29) | 7
  Harris Hip Function and Activity Score at 2 Years Subjects with a "Severe Dysfunction" Score (10-19): number analyzed (Participants) | 123
  Harris Hip Function and Activity Score at 2 Years Subjects with a "Severe Dysfunction" Score (10-19): number analyzed (Participant Hips) | 123
  Harris Hip Function and Activity Score at 2 Years Subjects with a "Severe Dysfunction" Score (10-19) | 1
  Harris Hip Function and Activity Score at 2 Years Subjects with a "Disabled" Score (0-9): number analyzed (Participants) | 123
  Harris Hip Function and Activity Score at 2 Years Subjects with a "Disabled" Score (0-9): number analyzed (Participant Hips) | 123
  Harris Hip Function and Activity Score at 2 Years Subjects with a "Disabled" Score (0-9) | 0
  Harris Hip Function and Activity Score at 3 Years Subjects with a "Normal" Score (40-47): number analyzed (Participants) | 67
  Harris Hip Function and Activity Score at 3 Years Subjects with a "Normal" Score (40-47): number analyzed (Participant Hips) | 67
  Harris Hip Function and Activity Score at 3 Years Subjects with a "Normal" Score (40-47) | 51
  Harris Hip Function and Activity Score at 3 Years Subjects with a "Mild Dysfunction" Score (30-39): number analyzed (Participants) | 67
  Harris Hip Function and Activity Score at 3 Years Subjects with a "Mild Dysfunction" Score (30-39): number analyzed (Participant Hips) | 67
  Harris Hip Function and Activity Score at 3 Years Subjects with a "Mild Dysfunction" Score (30-39) | 12
  Harris Hip Function and Activity Score at 3 Yrs Subjects with a "Moderate Dysfunction" Score (20-29): number analyzed (Participants) | 67
  Harris Hip Function and Activity Score at 3 Yrs Subjects with a "Moderate Dysfunction" Score (20-29): number analyzed (Participant Hips) | 67
  Harris Hip Function and Activity Score at 3 Yrs Subjects with a "Moderate Dysfunction" Score (20-29) | 3
  Harris Hip Function and Activity Score at 3 Years Subjects with a "Severe Dysfunction" Score (10-19): number analyzed (Participants) | 67
  Harris Hip Function and Activity Score at 3 Years Subjects with a "Severe Dysfunction" Score (10-19): number analyzed (Participant Hips) | 67
  Harris Hip Function and Activity Score at 3 Years Subjects with a "Severe Dysfunction" Score (10-19) | 1
  Harris Hip Function and Activity Score at 3 Years Subjects with a "Disabled" Score (0-9): number analyzed (Participants) | 67
  Harris Hip Function and Activity Score at 3 Years Subjects with a "Disabled" Score (0-9): number analyzed (Participant Hips) | 67
  Harris Hip Function and Activity Score at 3 Years Subjects with a "Disabled" Score (0-9) | 0
  Harris Hip Function and Activity Score at 4 Years Subjects with a "Normal" Score (40-47): number analyzed (Participants) | 35
  Harris Hip Function and Activity Score at 4 Years Subjects with a "Normal" Score (40-47): number analyzed (Participant Hips) | 35
  Harris Hip Function and Activity Score at 4 Years Subjects with a "Normal" Score (40-47) | 20
  Harris Hip Function and Activity Score at 4 Years Subjects with a "Mild Dysfunction" Score (30-39): number analyzed (Participants) | 35
  Harris Hip Function and Activity Score at 4 Years Subjects with a "Mild Dysfunction" Score (30-39): number analyzed (Participant Hips) | 35
  Harris Hip Function and Activity Score at 4 Years Subjects with a "Mild Dysfunction" Score (30-39) | 9
  Harris Hip Function and Activity Score at 4 Yrs Subjects with a "Moderate Dysfunction" Score (20-29): number analyzed (Participants) | 35
  Harris Hip Function and Activity Score at 4 Yrs Subjects with a "Moderate Dysfunction" Score (20-29): number analyzed (Participant Hips) | 35
  Harris Hip Function and Activity Score at 4 Yrs Subjects with a "Moderate Dysfunction" Score (20-29) | 5
  Harris Hip Function and Activity Score at 4 Years Subjects with a "Severe Dysfunction" Score (10-19): number analyzed (Participants) | 35
  Harris Hip Function and Activity Score at 4 Years Subjects with a "Severe Dysfunction" Score (10-19): number analyzed (Participant Hips) | 35
  Harris Hip Function and Activity Score at 4 Years Subjects with a "Severe Dysfunction" Score (10-19) | 0
  Harris Hip Function and Activity Score at 4 Years Subjects with a "Disabled" Score (0-9): number analyzed (Participants) | 35
  Harris Hip Function and Activity Score at 4 Years Subjects with a "Disabled" Score (0-9): number analyzed (Participant Hips) | 35
  Harris Hip Function and Activity Score at 4 Years Subjects with a "Disabled" Score (0-9) | 1
  Harris Hip Function and Activity Score at 5 Years Subjects with a "Normal" Score (40-47): number analyzed (Participants) | 110
  Harris Hip Function and Activity Score at 5 Years Subjects with a "Normal" Score (40-47): number analyzed (Participant Hips) | 110
  Harris Hip Function and Activity Score at 5 Years Subjects with a "Normal" Score (40-47) | 87
  Harris Hip Function and Activity Score at 5 Years Subjects with a "Mild Dysfunction" Score (30-39): number analyzed (Participants) | 110
  Harris Hip Function and Activity Score at 5 Years Subjects with a "Mild Dysfunction" Score (30-39): number analyzed (Participant Hips) | 110
  Harris Hip Function and Activity Score at 5 Years Subjects with a "Mild Dysfunction" Score (30-39) | 14
  Harris Hip Function and Activity Score at 5 Yrs Subjects with a "Moderate Dysfunction" Score (20-29): number analyzed (Participants) | 110
  Harris Hip Function and Activity Score at 5 Yrs Subjects with a "Moderate Dysfunction" Score (20-29): number analyzed (Participant Hips) | 110
  Harris Hip Function and Activity Score at 5 Yrs Subjects with a "Moderate Dysfunction" Score (20-29) | 6
  Harris Hip Function and Activity Score at 5 Years Subjects with a "Severe Dysfunction" Score (10-19): number analyzed (Participants) | 110
  Harris Hip Function and Activity Score at 5 Years Subjects with a "Severe Dysfunction" Score (10-19): number analyzed (Participant Hips) | 110
  Harris Hip Function and Activity Score at 5 Years Subjects with a "Severe Dysfunction" Score (10-19) | 2
  Harris Hip Function and Activity Score at 5 Years Subjects with a "Disabled" Score (0-9): number analyzed (Participants) | 110
  Harris Hip Function and Activity Score at 5 Years Subjects with a "Disabled" Score (0-9): number analyzed (Participant Hips) | 110
  Harris Hip Function and Activity Score at 5 Years Subjects with a "Disabled" Score (0-9) | 1

6. Secondary Outcome: Acetabular Cup Version - Annual Measurements
Description: Acetabular cup version is the angle formed between the axis of the implant and the coronal plane of the body. Acetabular version typically ranges between 11.5 and 28.5 degrees.
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Participant hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 107
Number analyzed (Participant hips) | 107
Degrees
  Acetabular cup version degrees, measured at 1 year | 22.8 (8.73)
  Acetabular cup version degrees, measured at 2 years: number analyzed (Participants) | 100
  Acetabular cup version degrees, measured at 2 years: number analyzed (Participant hips) | 100
  Acetabular cup version degrees, measured at 2 years | 23.7 (7.51)
  Acetabular cup version degrees, measured at 3 years: number analyzed (Participants) | 51
  Acetabular cup version degrees, measured at 3 years: number analyzed (Participant hips) | 51
  Acetabular cup version degrees, measured at 3 years | 25.1 (5.56)
  Acetabular cup version degrees, measured at 4 years: number analyzed (Participants) | 29
  Acetabular cup version degrees, measured at 4 years: number analyzed (Participant hips) | 29
  Acetabular cup version degrees, measured at 4 years | 23.8 (6.42)
  Acetabular cup version degrees, measured at 5 years: number analyzed (Participants) | 76
  Acetabular cup version degrees, measured at 5 years: number analyzed (Participant hips) | 76
  Acetabular cup version degrees, measured at 5 years | 26.1 (5.13)

7. Secondary Outcome: Acetabular Cup Inclination
Description: Acetabular cup inclination is the angle between the longitudinal axis of the patient and a perpendicular line to the major axis of the cup projection. The target acetabular cup inclination is between 30-50 degrees
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Participant Hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 124
Number analyzed (Participant Hips) | 124
Degrees
  Acetabular cup inclination, measured at 1 year | 42.9 (8.76)
  Acetabular cup inclination, measured at 2 years: number analyzed (Participants) | 120
  Acetabular cup inclination, measured at 2 years: number analyzed (Participant Hips) | 120
  Acetabular cup inclination, measured at 2 years | 42.2 (8.19)
  Acetabular cup inclination, measured at 3 years: number analyzed (Participants) | 66
  Acetabular cup inclination, measured at 3 years: number analyzed (Participant Hips) | 66
  Acetabular cup inclination, measured at 3 years | 42.6 (7.62)
  Acetabular cup inclination, measured at 4 years: number analyzed (Participants) | 32
  Acetabular cup inclination, measured at 4 years: number analyzed (Participant Hips) | 32
  Acetabular cup inclination, measured at 4 years | 43 (8.44)
  Acetabular cup inclination, measured at 5 years: number analyzed (Participants) | 107
  Acetabular cup inclination, measured at 5 years: number analyzed (Participant Hips) | 107
  Acetabular cup inclination, measured at 5 years | 43.5 (8.05)

8. Secondary Outcome: Acetabular Cup Migration
Description: Acetabular migration is the superior migration of the implant within the pelvic bone
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Count of Units; unit: Participant Hips
Units Other Than Participants: Participant Hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 126
Number analyzed (Participant Hips) | 126
Participant Hips
  Number of Participants with acetabular cup migration at 1 year | 0
  Number of Participants with acetabular cup migration at 2 years: number analyzed (Participants) | 124
  Number of Participants with acetabular cup migration at 2 years: number analyzed (Participant Hips) | 124
  Number of Participants with acetabular cup migration at 2 years | 0
  Number of Participants with acetabular cup migration at 3 years: number analyzed (Participants) | 66
  Number of Participants with acetabular cup migration at 3 years: number analyzed (Participant Hips) | 66
  Number of Participants with acetabular cup migration at 3 years | 0
  Number of Participants with acetabular cup migration at 4 years: number analyzed (Participants) | 35
  Number of Participants with acetabular cup migration at 4 years: number analyzed (Participant Hips) | 35
  Number of Participants with acetabular cup migration at 4 years | 0
  Number of Participants with acetabular cup migration at 5 years: number analyzed (Participants) | 109
  Number of Participants with acetabular cup migration at 5 years: number analyzed (Participant Hips) | 109
  Number of Participants with acetabular cup migration at 5 years | 0

9. Secondary Outcome: Heterotopic Ossification
Description: Heterotopic ossification is the abnormal formation of bone in soft tissues, such as muscles, tendons, or ligaments and can occur around the hip joint, leading to pain, stiffness, and restricted range of motion. It is graded as Class 0 through Class IV, with Class 0 being least impactful and Class IV being most impactful
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Count of Units; unit: Participant Hips
Units Other Than Participants: Participant Hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant Hips) | 127
Participant Hips
  Heterotopic Calcification at 1 year. Categories 0 - IV, and unable to assess: Class 0 | 87
  Heterotopic Calcification at 1 year. Categories 0 - IV, and unable to assess: Class I | 15
  Heterotopic Calcification at 1 year. Categories 0 - IV, and unable to assess: Class II | 21
  Heterotopic Calcification at 1 year. Categories 0 - IV, and unable to assess: Class III | 3
  Heterotopic Calcification at 1 year. Categories 0 - IV, and unable to assess: Class IV | 0
  Heterotopic Calcification at 1 year. Categories 0 - IV, and unable to assess: Unable to assess | 1
  Heterotopic Calcification at 2 years. Categories 0 - IV, and unable to assess: number analyzed (Participants) | 124
  Heterotopic Calcification at 2 years. Categories 0 - IV, and unable to assess: number analyzed (Participant Hips) | 124
  Heterotopic Calcification at 2 years. Categories 0 - IV, and unable to assess: Class 0 | 78
  Heterotopic Calcification at 2 years. Categories 0 - IV, and unable to assess: Class I | 17
  Heterotopic Calcification at 2 years. Categories 0 - IV, and unable to assess: Class II | 25
  Heterotopic Calcification at 2 years. Categories 0 - IV, and unable to assess: Class III | 4
  Heterotopic Calcification at 2 years. Categories 0 - IV, and unable to assess: Class IV | 0
  Heterotopic Calcification at 2 years. Categories 0 - IV, and unable to assess: Unable to assess | 0
  Heterotopic Calcification at 3 years. Categories 0 - IV, and unable to assess: number analyzed (Participants) | 66
  Heterotopic Calcification at 3 years. Categories 0 - IV, and unable to assess: number analyzed (Participant Hips) | 66
  Heterotopic Calcification at 3 years. Categories 0 - IV, and unable to assess: Class 0 | 32
  Heterotopic Calcification at 3 years. Categories 0 - IV, and unable to assess: Class I | 10
  Heterotopic Calcification at 3 years. Categories 0 - IV, and unable to assess: Class II | 22
  Heterotopic Calcification at 3 years. Categories 0 - IV, and unable to assess: Class III | 2
  Heterotopic Calcification at 3 years. Categories 0 - IV, and unable to assess: Class IV | 0
  Heterotopic Calcification at 3 years. Categories 0 - IV, and unable to assess: Unable to assess | 0
  Heterotopic Calcification at 4 years. Categories 0 - IV, and unable to assess: number analyzed (Participants) | 35
  Heterotopic Calcification at 4 years. Categories 0 - IV, and unable to assess: number analyzed (Participant Hips) | 35
  Heterotopic Calcification at 4 years. Categories 0 - IV, and unable to assess: Class 0 | 21
  Heterotopic Calcification at 4 years. Categories 0 - IV, and unable to assess: Class I | 5
  Heterotopic Calcification at 4 years. Categories 0 - IV, and unable to assess: Class II | 7
  Heterotopic Calcification at 4 years. Categories 0 - IV, and unable to assess: Class III | 2
  Heterotopic Calcification at 4 years. Categories 0 - IV, and unable to assess: Class IV | 0
  Heterotopic Calcification at 4 years. Categories 0 - IV, and unable to assess: Unable to assess | 0
  Heterotopic Calcification at 5 years. Categories 0 - IV, and unable to assess: number analyzed (Participants) | 109
  Heterotopic Calcification at 5 years. Categories 0 - IV, and unable to assess: number analyzed (Participant Hips) | 109
  Heterotopic Calcification at 5 years. Categories 0 - IV, and unable to assess: Class 0 | 64
  Heterotopic Calcification at 5 years. Categories 0 - IV, and unable to assess: Class I | 16
  Heterotopic Calcification at 5 years. Categories 0 - IV, and unable to assess: Class II | 26
  Heterotopic Calcification at 5 years. Categories 0 - IV, and unable to assess: Class III | 3
  Heterotopic Calcification at 5 years. Categories 0 - IV, and unable to assess: Class IV | 0
  Heterotopic Calcification at 5 years. Categories 0 - IV, and unable to assess: Unable to assess | 0

10. Secondary Outcome: Acetabular Radiolucent Lines
Description: Radiolucent lines are seen on x-rays and represent an area that is absent of bone. Radiolucent lines seen adjacent to an implant may suggest a lack on bone ingrowth or possible loosening of the implant.
  Radiolucent lines greater than 1mm wide were considered reportable for this study.
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Count of Units; unit: Participant hips
Units Other Than Participants: Participant hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant hips) | 127
Participant hips
  Number of study Participants with radiolucent lines greater than 1mm in width at 1 year | 1
  Number of study Participants with radiolucent lines greater than 1mm in width at 2 years: number analyzed (Participants) | 124
  Number of study Participants with radiolucent lines greater than 1mm in width at 2 years: number analyzed (Participant hips) | 124
  Number of study Participants with radiolucent lines greater than 1mm in width at 2 years | 1
  Number of study Participants with radiolucent lines greater than 1mm in width at 3 years: number analyzed (Participants) | 66
  Number of study Participants with radiolucent lines greater than 1mm in width at 3 years: number analyzed (Participant hips) | 66
  Number of study Participants with radiolucent lines greater than 1mm in width at 3 years | 1
  Number of study Participants with radiolucent lines greater than 1mm in width at 4 years: number analyzed (Participants) | 35
  Number of study Participants with radiolucent lines greater than 1mm in width at 4 years: number analyzed (Participant hips) | 35
  Number of study Participants with radiolucent lines greater than 1mm in width at 4 years | 1
  Number of study Participants with radiolucent lines greater than 1mm in width at 5 years: number analyzed (Participants) | 109
  Number of study Participants with radiolucent lines greater than 1mm in width at 5 years: number analyzed (Participant hips) | 109
  Number of study Participants with radiolucent lines greater than 1mm in width at 5 years | 1

11. Secondary Outcome: Acetabular Osteolysis
Description: Osteolysis is seen on x-rays and represent an area where bone has been resorbed by the body in response to small particles of debris that are created as an implant wears over time. Osteolysis greater than 5mm was considered to be reportable for this study.
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Count of Units; unit: Participant hips
Units Other Than Participants: Participant hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant hips) | 127
Participant hips
  Number of study Participants with acetabular osteolysis at 1 year | 2
  Number of study Participants with acetabular osteolysis at 2 years: number analyzed (Participants) | 124
  Number of study Participants with acetabular osteolysis at 2 years: number analyzed (Participant hips) | 124
  Number of study Participants with acetabular osteolysis at 2 years | 2
  Number of study Participants with acetabular osteolysis at 3 years: number analyzed (Participants) | 66
  Number of study Participants with acetabular osteolysis at 3 years: number analyzed (Participant hips) | 66
  Number of study Participants with acetabular osteolysis at 3 years | 0
  Number of study Participants with acetabular osteolysis at 4 years: number analyzed (Participants) | 35
  Number of study Participants with acetabular osteolysis at 4 years: number analyzed (Participant hips) | 35
  Number of study Participants with acetabular osteolysis at 4 years | 0
  Number of study Participants with acetabular osteolysis at 5 years: number analyzed (Participants) | 109
  Number of study Participants with acetabular osteolysis at 5 years: number analyzed (Participant hips) | 109
  Number of study Participants with acetabular osteolysis at 5 years | 1

12. Secondary Outcome: Acetabular Sclerotic Lines
Description: Acetabular sclerotic lines are seen on x-rays and are radio-dense areas of bone that have remodeled due to loads close to the implant.
Time Frame: Measured from x-rays taken annually, years 1 though 5
Population: All study participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Count of Units; unit: Participant Hips
Units Other Than Participants: Participant Hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant Hips) | 127
Participant Hips
  Number of study Participants with acetabular sclerotic lines present at 1 Year | 1
  Number of study Participants with acetabular sclerotic lines present at 2 Years: number analyzed (Participants) | 124
  Number of study Participants with acetabular sclerotic lines present at 2 Years: number analyzed (Participant Hips) | 124
  Number of study Participants with acetabular sclerotic lines present at 2 Years | 3
  Number of study Participants with acetabular sclerotic lines present at 3 Years: number analyzed (Participants) | 66
  Number of study Participants with acetabular sclerotic lines present at 3 Years: number analyzed (Participant Hips) | 66
  Number of study Participants with acetabular sclerotic lines present at 3 Years | 3
  Number of study Participants with acetabular sclerotic lines present at 4 Years: number analyzed (Participants) | 35
  Number of study Participants with acetabular sclerotic lines present at 4 Years: number analyzed (Participant Hips) | 35
  Number of study Participants with acetabular sclerotic lines present at 4 Years | 3
  Number of study Participants with acetabular sclerotic lines present at 5 Years: number analyzed (Participants) | 109
  Number of study Participants with acetabular sclerotic lines present at 5 Years: number analyzed (Participant Hips) | 109
  Number of study Participants with acetabular sclerotic lines present at 5 Years | 3

13. Secondary Outcome: Femoral Stem Position
Description: Femoral stem position is categorized as neutral, valgus, or varus. A neutral stem is centered within the femoral canal that runs through the center of the femur's long axis. A valgus femoral stem is positioned slightly towards the medial side of the femoral canal, and a varus femoral stem is positioned slightly towards the lateral side of the femoral canal.
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Count of Units; unit: Participant hips
Units Other Than Participants: Participant hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant hips) | 127
Participant hips
  Femoral stem position in study patients at 1 year follow-up: Number with Neutral stem position | 79
  Femoral stem position in study patients at 1 year follow-up: Number with Valgus stem position | 10
  Femoral stem position in study patients at 1 year follow-up: Number with Varus stem position | 35
  Femoral stem position in study patients at 1 year follow-up: Unable to assess | 2
  Femoral stem position in study patients at 1 year follow-up: Indeterminate | 1
  Femoral stem position in study patients at 2 year follow-up: number analyzed (Participants) | 124
  Femoral stem position in study patients at 2 year follow-up: number analyzed (Participant hips) | 124
  Femoral stem position in study patients at 2 year follow-up: Number with Neutral stem position | 77
  Femoral stem position in study patients at 2 year follow-up: Number with Valgus stem position | 9
  Femoral stem position in study patients at 2 year follow-up: Number with Varus stem position | 38
  Femoral stem position in study patients at 2 year follow-up: Unable to assess | 0
  Femoral stem position in study patients at 2 year follow-up: Indeterminate | 0
  Femoral stem position in study patients at 3 year follow-up: number analyzed (Participants) | 66
  Femoral stem position in study patients at 3 year follow-up: number analyzed (Participant hips) | 66
  Femoral stem position in study patients at 3 year follow-up: Number with Neutral stem position | 35
  Femoral stem position in study patients at 3 year follow-up: Number with Valgus stem position | 6
  Femoral stem position in study patients at 3 year follow-up: Number with Varus stem position | 24
  Femoral stem position in study patients at 3 year follow-up: Unable to assess | 1
  Femoral stem position in study patients at 3 year follow-up: Indeterminate | 0
  Femoral stem position in study patients at 4 year follow-up: number analyzed (Participants) | 35
  Femoral stem position in study patients at 4 year follow-up: number analyzed (Participant hips) | 35
  Femoral stem position in study patients at 4 year follow-up: Number with Neutral stem position | 19
  Femoral stem position in study patients at 4 year follow-up: Number with Valgus stem position | 4
  Femoral stem position in study patients at 4 year follow-up: Number with Varus stem position | 12
  Femoral stem position in study patients at 4 year follow-up: Unable to assess | 0
  Femoral stem position in study patients at 4 year follow-up: Indeterminate | 0
  Femoral stem position in study patients at 5 year follow-up: number analyzed (Participants) | 109
  Femoral stem position in study patients at 5 year follow-up: number analyzed (Participant hips) | 109
  Femoral stem position in study patients at 5 year follow-up: Number with Neutral stem position | 67
  Femoral stem position in study patients at 5 year follow-up: Number with Valgus stem position | 8
  Femoral stem position in study patients at 5 year follow-up: Number with Varus stem position | 34
  Femoral stem position in study patients at 5 year follow-up: Unable to assess | 0
  Femoral stem position in study patients at 5 year follow-up: Indeterminate | 0

14. Secondary Outcome: Femoral Stem Tilt
Description: Femoral stem tilt is a measurement taken at each post-operative year and compared against baseline images collected at 6-weeks post-operative. The measurement captures changes in the position of the femoral stem over time. Tilt greater than 2 degrees was considered reportable for this study
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Count of Units; unit: Participant hips
Units Other Than Participants: Participant hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant hips) | 127
Participant hips
  Number of Study Participants with femoral tilt greater than 2 degrees at 1 year | 3
  Number of Study Participants with femoral tilt greater than 2 degrees at 2 years: number analyzed (Participants) | 124
  Number of Study Participants with femoral tilt greater than 2 degrees at 2 years: number analyzed (Participant hips) | 124
  Number of Study Participants with femoral tilt greater than 2 degrees at 2 years | 3
  Number of Study Participants with femoral tilt greater than 2 degrees at 3 years: number analyzed (Participants) | 66
  Number of Study Participants with femoral tilt greater than 2 degrees at 3 years: number analyzed (Participant hips) | 66
  Number of Study Participants with femoral tilt greater than 2 degrees at 3 years | 3
  Number of Study Participants with femoral tilt greater than 2 degrees at 4 years: number analyzed (Participants) | 35
  Number of Study Participants with femoral tilt greater than 2 degrees at 4 years: number analyzed (Participant hips) | 35
  Number of Study Participants with femoral tilt greater than 2 degrees at 4 years | 2
  Number of Study Participants with femoral tilt greater than 2 degrees at 5 years: number analyzed (Participants) | 109
  Number of Study Participants with femoral tilt greater than 2 degrees at 5 years: number analyzed (Participant hips) | 109
  Number of Study Participants with femoral tilt greater than 2 degrees at 5 years | 5

15. Secondary Outcome: Femoral Stem Subsidence
Description: Femoral stem subsidence is the inferior movement of the stem within the femoral canal. Subsidence greater than 2 mm was considered reportable for this study.
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Count of Units; unit: Participant hips
Units Other Than Participants: Participant hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant hips) | 127
Participant hips
  Number of study Participants with femoral stem subsidence greater that 2mm at 1 year | 0
  Number of study Participants with femoral stem subsidence greater that 2mm at 2 years: number analyzed (Participants) | 124
  Number of study Participants with femoral stem subsidence greater that 2mm at 2 years: number analyzed (Participant hips) | 124
  Number of study Participants with femoral stem subsidence greater that 2mm at 2 years | 0
  Number of study Participants with femoral stem subsidence greater that 2mm at 3 years: number analyzed (Participants) | 66
  Number of study Participants with femoral stem subsidence greater that 2mm at 3 years: number analyzed (Participant hips) | 66
  Number of study Participants with femoral stem subsidence greater that 2mm at 3 years | 0
  Number of study Participants with femoral stem subsidence greater that 2mm at 4 years: number analyzed (Participants) | 35
  Number of study Participants with femoral stem subsidence greater that 2mm at 4 years: number analyzed (Participant hips) | 35
  Number of study Participants with femoral stem subsidence greater that 2mm at 4 years | 0
  Number of study Participants with femoral stem subsidence greater that 2mm at 5 years: number analyzed (Participants) | 109
  Number of study Participants with femoral stem subsidence greater that 2mm at 5 years: number analyzed (Participant hips) | 109
  Number of study Participants with femoral stem subsidence greater that 2mm at 5 years | 0

16. Secondary Outcome: Femoral Stem Heterotopic Ossification
Description: Heterotopic ossification is the abnormal formation of bone in soft tissues such as muscles, tendons, or ligaments and can occur around the hip joint, leading to pain, stiffness, and restricted range of motion. It is graded as Class 0 through Class IV, with Class O having no bone growth in soft tissue, Class I being least impactful and Class IV being most impactful.
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study Participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Count of Units; unit: Participant hips
Units Other Than Participants: Participant hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant hips) | 127
Participant hips
  Study Participant Femoral Heterotopic Ossification at 1 year: Class 0 | 87
  Study Participant Femoral Heterotopic Ossification at 1 year: Class I | 21
  Study Participant Femoral Heterotopic Ossification at 1 year: Class II | 14
  Study Participant Femoral Heterotopic Ossification at 1 year: Class III | 3
  Study Participant Femoral Heterotopic Ossification at 1 year: Class IV | 0
  Study Participant Femoral Heterotopic Ossification at 1 year: Unable to assess | 2
  Study Participant Femoral Heterotopic Ossification at 2 years: number analyzed (Participants) | 124
  Study Participant Femoral Heterotopic Ossification at 2 years: number analyzed (Participant hips) | 124
  Study Participant Femoral Heterotopic Ossification at 2 years: Class 0 | 80
  Study Participant Femoral Heterotopic Ossification at 2 years: Class I | 21
  Study Participant Femoral Heterotopic Ossification at 2 years: Class II | 17
  Study Participant Femoral Heterotopic Ossification at 2 years: Class III | 6
  Study Participant Femoral Heterotopic Ossification at 2 years: Class IV | 0
  Study Participant Femoral Heterotopic Ossification at 2 years: Unable to assess | 0
  Study Participant Femoral Heterotopic Ossification at 3 years: number analyzed (Participants) | 66
  Study Participant Femoral Heterotopic Ossification at 3 years: number analyzed (Participant hips) | 66
  Study Participant Femoral Heterotopic Ossification at 3 years: Class 0 | 40
  Study Participant Femoral Heterotopic Ossification at 3 years: Class I | 13
  Study Participant Femoral Heterotopic Ossification at 3 years: Class II | 10
  Study Participant Femoral Heterotopic Ossification at 3 years: Class III | 3
  Study Participant Femoral Heterotopic Ossification at 3 years: Class IV | 0
  Study Participant Femoral Heterotopic Ossification at 3 years: Unable to assess | 0
  Study Participant Femoral Heterotopic Ossification at 4 years: number analyzed (Participants) | 35
  Study Participant Femoral Heterotopic Ossification at 4 years: number analyzed (Participant hips) | 35
  Study Participant Femoral Heterotopic Ossification at 4 years: Class 0 | 21
  Study Participant Femoral Heterotopic Ossification at 4 years: Class I | 8
  Study Participant Femoral Heterotopic Ossification at 4 years: Class II | 3
  Study Participant Femoral Heterotopic Ossification at 4 years: Class III | 3
  Study Participant Femoral Heterotopic Ossification at 4 years: Class IV | 0
  Study Participant Femoral Heterotopic Ossification at 4 years: Unable to assess | 0
  Study Participant Femoral Heterotopic Ossification at 5 years: number analyzed (Participants) | 109
  Study Participant Femoral Heterotopic Ossification at 5 years: number analyzed (Participant hips) | 109
  Study Participant Femoral Heterotopic Ossification at 5 years: Class 0 | 65
  Study Participant Femoral Heterotopic Ossification at 5 years: Class I | 21
  Study Participant Femoral Heterotopic Ossification at 5 years: Class II | 19
  Study Participant Femoral Heterotopic Ossification at 5 years: Class III | 4
  Study Participant Femoral Heterotopic Ossification at 5 years: Class IV | 0
  Study Participant Femoral Heterotopic Ossification at 5 years: Unable to assess | 0

17. Secondary Outcome: Femoral Radiolucent Lines
Description: Radiolucencies are seen on x-rays and represent an area that is absent of bone. Radiolucent lines seen adjacent to an implant may suggest a lack of bone ingrowth into the implant or possible loosening of the implant
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study Participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Number; unit: Participants
Units Other Than Participants: Participant Hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant Hips) | 127
Participants
  Study Participants with femoral radiolucent lines present at 1 year | 0
  Study Participants with femoral radiolucent lines present at 2 years: number analyzed (Participants) | 124
  Study Participants with femoral radiolucent lines present at 2 years: number analyzed (Participant Hips) | 124
  Study Participants with femoral radiolucent lines present at 2 years | 1
  Study Participants with femoral radiolucent lines present at 3 years: number analyzed (Participants) | 66
  Study Participants with femoral radiolucent lines present at 3 years: number analyzed (Participant Hips) | 66
  Study Participants with femoral radiolucent lines present at 3 years | 0
  Study Participants with femoral radiolucent lines present at 4 years: number analyzed (Participants) | 35
  Study Participants with femoral radiolucent lines present at 4 years: number analyzed (Participant Hips) | 35
  Study Participants with femoral radiolucent lines present at 4 years | 0
  Study Participants with femoral radiolucent lines present at 5 years: number analyzed (Participants) | 109
  Study Participants with femoral radiolucent lines present at 5 years: number analyzed (Participant Hips) | 109
  Study Participants with femoral radiolucent lines present at 5 years | 0

18. Secondary Outcome: Femoral Osteolysis
Description: as for outcome 11
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study Participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Number; unit: Participants
Units Other Than Participants: Participant Hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant Hips) | 127
Participants
  Number of study Participants with femoral osteolysis at 1 year | 0
  Number of study Participants with femoral osteolysis at 2 years: number analyzed (Participants) | 124
  Number of study Participants with femoral osteolysis at 2 years: number analyzed (Participant Hips) | 124
  Number of study Participants with femoral osteolysis at 2 years | 0
  Number of study Participants with femoral osteolysis at 3 years: number analyzed (Participants) | 66
  Number of study Participants with femoral osteolysis at 3 years: number analyzed (Participant Hips) | 66
  Number of study Participants with femoral osteolysis at 3 years | 0
  Number of study Participants with femoral osteolysis at 4 years: number analyzed (Participants) | 35
  Number of study Participants with femoral osteolysis at 4 years: number analyzed (Participant Hips) | 35
  Number of study Participants with femoral osteolysis at 4 years | 0
  Number of study Participants with femoral osteolysis at 5 years: number analyzed (Participants) | 109
  Number of study Participants with femoral osteolysis at 5 years: number analyzed (Participant Hips) | 109
  Number of study Participants with femoral osteolysis at 5 years | 0

19. Secondary Outcome: Femoral Stem Sclerotic Lines
Description: as for outcome 12
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study Participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Number; unit: Participants
Units Other Than Participants: Participant Hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant Hips) | 127
Participants
  Number of study participants with femoral sclerotic lines present at 1 year | 1
  Number of study participants with femoral sclerotic lines present at 2 years: number analyzed (Participants) | 124
  Number of study participants with femoral sclerotic lines present at 2 years: number analyzed (Participant Hips) | 124
  Number of study participants with femoral sclerotic lines present at 2 years | 5
  Number of study participants with femoral sclerotic lines present at 3 years: number analyzed (Participants) | 66
  Number of study participants with femoral sclerotic lines present at 3 years: number analyzed (Participant Hips) | 66
  Number of study participants with femoral sclerotic lines present at 3 years | 5
  Number of study participants with femoral sclerotic lines present at 4 years: number analyzed (Participants) | 35
  Number of study participants with femoral sclerotic lines present at 4 years: number analyzed (Participant Hips) | 35
  Number of study participants with femoral sclerotic lines present at 4 years | 1
  Number of study participants with femoral sclerotic lines present at 5 years: number analyzed (Participants) | 109
  Number of study participants with femoral sclerotic lines present at 5 years: number analyzed (Participant Hips) | 109
  Number of study participants with femoral sclerotic lines present at 5 years | 7

20. Secondary Outcome: Femoral Stem Calcar Resorption
Description: Femoral calcar resorption occurs when the bone around the prosthesis is partially shielded from bearing loads and begins to resorb
Time Frame: Measure from x-rays taken annually, years 1 through 5
Population: All study Participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Number; unit: Participants
Units Other Than Participants: Participant Hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant Hips) | 127
Participants
  Study patients with calcar resorption indicated on x-rays at 1 year | 1
  Study patients with calcar resorption indicated on x-rays at 2 years: number analyzed (Participants) | 124
  Study patients with calcar resorption indicated on x-rays at 2 years: number analyzed (Participant Hips) | 124
  Study patients with calcar resorption indicated on x-rays at 2 years | 2
  Study patients with calcar resorption indicated on x-rays at 3 years: number analyzed (Participants) | 66
  Study patients with calcar resorption indicated on x-rays at 3 years: number analyzed (Participant Hips) | 66
  Study patients with calcar resorption indicated on x-rays at 3 years | 2
  Study patients with calcar resorption indicated on x-rays at 4 years: number analyzed (Participants) | 35
  Study patients with calcar resorption indicated on x-rays at 4 years: number analyzed (Participant Hips) | 35
  Study patients with calcar resorption indicated on x-rays at 4 years | 2
  Study patients with calcar resorption indicated on x-rays at 5 years: number analyzed (Participants) | 109
  Study patients with calcar resorption indicated on x-rays at 5 years: number analyzed (Participant Hips) | 109
  Study patients with calcar resorption indicated on x-rays at 5 years | 3

21. Secondary Outcome: Femoral Stem Calcar Fracture
Description: Near the top of the femur is a region of bone called the calcar femorale that provides strength to the femur when compressive forces are applied. During preparation of the femur to receive the femoral implant there is the possibility of fractures occurring in this region
Time Frame: Measured from x-rays taken annually, years 1 through 5
Population: All study Participants who returned for scheduled follow-up clinic visits and had radiographic images taken
Measure: Number; unit: Participants
Units Other Than Participants: Participant hips
Arm/Group | CERAMAX COC 36mm Acetabular Cup
Number analyzed (Participants) | 127
Number analyzed (Participant hips) | 127
Participants
  Number of Study participants with a calcar fracture noted on x-rays at 1 year | 0
  Number of Study participants with a calcar fracture noted on x-rays at 2 years: number analyzed (Participants) | 124
  Number of Study participants with a calcar fracture noted on x-rays at 2 years: number analyzed (Participant hips) | 124
  Number of Study participants with a calcar fracture noted on x-rays at 2 years | 0
  Number of Study participants with a calcar fracture noted on x-rays at 3 years: number analyzed (Participants) | 66
  Number of Study participants with a calcar fracture noted on x-rays at 3 years: number analyzed (Participant hips) | 66
  Number of Study participants with a calcar fracture noted on x-rays at 3 years | 0
  Number of Study participants with a calcar fracture noted on x-rays at 4 years: number analyzed (Participants) | 35
  Number of Study participants with a calcar fracture noted on x-rays at 4 years: number analyzed (Participant hips) | 35
  Number of Study participants with a calcar fracture noted on x-rays at 4 years | 0
  Number of Study participants with a calcar fracture noted on x-rays at 5 years: number analyzed (Participants) | 109
  Number of Study participants with a calcar fracture noted on x-rays at 5 years: number analyzed (Participant hips) | 109
  Number of Study participants with a calcar fracture noted on x-rays at 5 years | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the course of the study and continued until the 5-year interval when the study closed
Description: Adverse events were collected throughout the course of the study and continued until the 5-year interval when the study closed
Arm/Group | CERAMAX COC 36mm Acetabular Cup
All-Cause Mortality (participants affected / at risk) | 2/170
Serious Adverse Events (participants affected / at risk) | 86/170
Other Adverse Events (participants affected / at risk) | 141/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CERAMAX COC 36mm Acetabular Cup (N=170)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (4)
Atrial flutter (Cardiac disorders) | 1 (4)
Coronary artery disease (Cardiac disorders) | 2 (2)
Foetal heart rate deceleration abnormality (Cardiac disorders) | 1 (1)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Anal stenosis (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (3)
Arthritis infective (Infections and infestations) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Empyema (Infections and infestations) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Medical device site joint infection (Infections and infestations) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Sepsis (Infections and infestations) | 2 (3)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 3 (3)
Joint effusion (Injury, poisoning and procedural complications) | 1 (2)
Joint instability (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 39 (39)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 7 (7)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2)
Synovial disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Alcoholic seizure (Nervous system disorders) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (2)
Device failure (Product Issues) | 2 (3)
Device loosening (Product Issues) | 3 (3)
Delirium tremens (Psychiatric disorders) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (11)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CERAMAX COC 36mm Acetabular Cup (N=170)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 37 (52)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 37 (48)
Bursitis (Musculoskeletal and connective tissue disorders) | 30 (35)
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 (29)
Back Pain (Musculoskeletal and connective tissue disorders) | 20 (24)
Fall (Injury, poisoning and procedural complications) | 19 (23)
Tendonitis (Musculoskeletal and connective tissue disorders) | 15 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (11)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT02096211/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT02096211/SAP_001.pdf